CLINICAL TRIAL: NCT06556082
Title: The Effect of Proprioceptive Neuromuscular Facilitation Based Upper Extremity Strengthening Exercises Combined With Core Stabilization Training on Physical Fitness Parameters in Amputee Football Players
Brief Title: Effect of PNF-Based Upper Extremity Strengthening With Core Stabilization on Fitness in Amputee Football Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Mert İlhan, MSc, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-RCTILHAN-01
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Amputation; Lower Limb Amputation
Keywords: Amputee Football; Physical Fitness; Balance
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Training and Control Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): In addition to the standard training programs in the off-season period; PNF-based upper extremity strengthening training will be performed 3 days a week for 8 weeks in addition to core stabilization training.
  Interventions: Other: Training
- Control Group (Experimental): The amputee football players in the control group will be trained 3 days a week for 8 weeks with isotonic strengthening exercises of the upper extremity muscles with free weights and core stabilization training.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Training — Proprioceptive Neuromuscular Facilitation(PNF) based upper extremity strengthening exercises to increase upper extremity muscle strength will be applied to the participants in the training group 3 days a week for 8 weeks. PNF-based upper extremity strengthening exercises will be performed with an elastic resistive band using bilateral symmetrical PNF patterns of "Flexion-Adduction-External Rotation-Extension-Abduction-Internal Rotation", "Flexion-Abduction-External Rotation-Extension-Adduction-Internal Rotation" on two different diagonals while individuals are in a sitting position in a supported chair. Core Stabilization Training will be continued for 8 weeks by increasing the difficulty and intensity of the exercises with limb movements and floor modifications after the amputee football players are taught how to find their neutral spine and how to maintain the position.
  Arms: Training Group
Other: Control Group — The control group will be trained with isotonic strengthening exercises of upper extremity muscles with free weights and core stabilization training 3 days a week for 8 weeks. Isotonic exercises involve muscle contraction with movement, where the muscle length changes while maintaining constant tension. Free weights such as dumbells will be used in the implementation of the exercises. 1 Repetition Maximum (1RM) method will be used to determine the progression of the exercises.
  Arms: Control Group

SUMMARY:
Amputee football (AF) is a disability-specific football in which amputees can participate. This study aims to determine the effect of PNF-based upper extremity strengthening exercises combined with core stabilization exercises on physical fitness parameters in amputee football players. In the study, amputee soccer players will be randomly divided into two groups training and control groups. In addition to the standard training programs in the off-season, the amputee athletes in the training group will receive PNF-based upper extremity strengthening training combined with core stabilization training by the same physiotherapist 3 days a week for 8 weeks. The amputee football players in the control group will be given upper extremity strengthening training with free weights in addition to core stabilization training 3 days a week for 8 weeks. The physical and demographic characteristics of the cases who signed the consent form will be recorded. Initial evaluations will be made before the start of the exercise training program and secondary evaluations will be made at the end of 8 weeks. Detailed information about the participants will be obtained with the Descriptive Characteristics Information Form. Single Leg Balance Test, Berg Balance Scale and Activity Specific Balance Confidence Scale will be used to obtain information about postural control and balance strategies of the participants. Pressure Feedback Unit will be used to measure the stabilization capacity of deep spinal muscles. Trunk muscle endurance tests developed by McGill will be used to assess the level of core stability. Isokinetic muscle strength of the upper extremity muscles will be measured with the ISOMED 2000 (2017-Germany) device. Hand grip strength will be measured with Jamar Hand Dynanometer. Closed Kinetic Ring Upper Extremity Test will be used to measure the strength, anaerobic power, and closed kinetic chain stability of the upper extremity. The Distance Triple Hop Test will be used to assess the strength, speed, balance, and control ability of a lower extremity with special emphasis on the distance traveled by the lower extremity. Sprint Test will be used to measure the running performance of amputee soccer players. The data will then be analyzed and interpreted with appropriate statistical methods.

DETAILED DESCRIPTION:
Amputee football (AF) is a disability-specific football in which amputees can participate. Optimum flexibility, strength, endurance, speed, and agility are required to perform adequately in amputee football. However, amputee soccer requires intense strength and stability requirements on the upper extremities and trunk, especially due to the use of crutches. The aim of this study is to determine the effect of PNF-based upper extremity strengthening exercises combined with core stabilization exercises on physical fitness parameters in amputee football players. In the study, amputee soccer players will be randomly divided into two groups training and control groups. In addition to the standard training programs in the off-season, the amputee athletes in the training group will receive PNF-based upper extremity strengthening training combined with core stabilization training by the same physiotherapist 3 days a week for 8 weeks. The amputee football players in the control group will be given upper extremity strengthening training with free weights in addition to core stabilization training 3 days a week for 8 weeks. The physical and demographic characteristics of the cases who signed the consent form will be recorded. Initial evaluations will be made before the start of the exercise training program and secondary evaluations will be made at the end of 8 weeks. Detailed information about the participants will be obtained with the Descriptive Characteristics Information Form. Single Leg Balance Test, Berg Balance Scale, and Activity Specific Balance Confidence Scale will be used to obtain information about postural control and balance strategies of the participants. Pressure Feedback Unit will be used to measure the stabilization capacity of deep spinal muscles. Trunk muscle endurance tests developed by McGill will be used to assess the level of core stability. Isokinetic muscle strength of the upper extremity muscles will be measured with the ISOMED 2000 (2017-Germany) device. Hand grip strength will be measured with Jamar Hand Dynanometer. Closed Kinetic Ring Upper Extremity Test will be used to measure the strength, anaerobic power, and closed kinetic chain stability of the upper extremity. The Distance Triple Hop Test will be used to assess the strength, speed, balance, and control ability of a lower extremity with special emphasis on the distance traveled by the lower extremity. Sprint Test will be used to measure the running performance of amputee soccer players. The data will then be analyzed and interpreted with appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* At least one year of experience in playing amputee soccer.
* Transtibial, knee disarticulation, or transfemoral level amputation.

Exclusion Criteria:

* Presence of upper extremity amputation.
* Bilateral lower extremity amputation.
* Underwent upper or lower extremity surgery within the last 6 months.
* Neurological disease, vestibular or visual problems.
* Use of medication affecting the central nervous system.
* Any pathology that may affect motor performance.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Isokinetic Upper Extremity Muscle Strength | Baseline (pre-intervention) and at 8 weeks (post-intervention).
  The strength of the shoulder, elbow, and wrist muscles will be assessed using an isokinetic dynamometer (ISOMED 2000). Measurements will be taken at angular velocities of 60°/s and 180°/s in concentric-concentric mode for abduction-adduction and internal-external rotation movements. The peak torque values will be recorded.
Core Muscle Strength | Baseline (pre-intervention) and at 8 weeks (post-intervention).
  Core muscle strength will be measured using the Stabilizer Pressure Biofeedback Unit (Chattanoga Group,2005). The device will be used to assess the ability of participants to maintain a neutral spine position during various core stabilization exercises.
Sprint Performance | Baseline (pre-intervention) and at 8 weeks (post-intervention).
  Sprint performance will be assessed by recording the time it takes for participants to complete 10m, 20m, and 30m sprints using crutches. Two trials will be conducted, and the best times will be recorded.

SECONDARY OUTCOMES:
Postural Stability | Baseline (pre-intervention) and at 8 weeks (post-intervention).
  The Berg Balance Scale will be used to assess the overall postural stability and balance of the participants. This test consists of 14 tasks that measure a range of balance activities, each scored from 0 to 4. Higher scores indicate better balance and stability.
Balance Confidence | Baseline (pre-intervention) and at 8 weeks (post-intervention).
  Activities-Specific Balance Confidence Scale (ABC) will assess the participants' confidence in maintaining balance during various activities. It includes 16 items scored from 0% (no confidence) to 100% (full confidence).
Static Balance Assessment | Baseline (pre-intervention) and at 8 weeks (post-intervention).
  The Single Leg Stance Test will be used to assess static balance and postural control. Participants will be asked to stand on one leg with their arms either on their hips or crossed over their shoulders. The time (in seconds) they can maintain balance without losing posture will be recorded. The best of three trials will be used for analysis.
Upper Extremity Endurance and Stability | Baseline (pre-intervention) and at 8 weeks (post-intervention).
  Closed Kinetic Chain Upper Extremity Stability Test will be used to assess upper extremity stability and endurance. Participants will perform in push-up position, touching two lines placed 0.9 meters apart as many times as possible within 15 seconds. The total number of touches will be recorded.
Grip Strength Assessment | Baseline (pre-intervention) and at 8 weeks (post-intervention).
  Grip strength will be measured using a Jamar hand dynamometer according to the American Society of Hand Therapists (ASHT) protocol. Participants will perform three trials with their dominant hand, and the average value will be recorded.
Athletic Performance (Triple Hop Distance Test) | Baseline (pre-intervention) and at 8 weeks (post-intervention).
  The Triple Hop Distance Test will be used to assess the explosive power, balance, and control of the lower extremity. Participants will be asked to hop as far as possible on one leg, three consecutive times without losing balance. The distance from the starting point to the final landing point will be measured and recorded.
Core Stability Level | Baseline (pre-intervention) and at 8 weeks (post-intervention).
  Core stability will be evaluated using the McGill core tests, which include the Sorensen test, trunk flexion test, and side bridge tests. These tests measure the endurance of the core muscles by recording the time (in seconds) participants can maintain specific postures.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Erbahçeci, PhD., Study Director — Hacettepe University
Locations (1):
- Uskudar University Physiotherapy and Rehabilitation Application and Research Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No